# Assessing Engagement Patterns and Participation Trends in Individuals Joining Anorexia Clinical Trials: An Observational Investigation

This is an Informed Consent Form For Anorexia Clinical Patients in <a href="Power Clinical Trial's">Power Clinical Trial's</a> Observational Study

Date: November 17, 2023

Overview of the Informed Consent Form for Potential Participants

Completing this form implies potential eligibility for involvement in a distinctive observational clinical investigation aimed at individuals dealing with anorexia. This comprehensive document outlines the study's fundamental objectives, the methodology employed, and the potential impacts, encompassing both positive and potentially adverse effects. Before deciding, it's crucial to thoroughly understand the potential implications of participation, and seeking guidance from your healthcare provider can offer valuable insights. If any part of this material seems unclear or if questions arise, please reach out to the researcher or the appointed contact person.

Significance of Clinical Trials in Addressing Anorexia

Clinical trials centered on anorexia serve a pivotal function in assessing the safety and effectiveness of emerging treatments for this condition. These trials stand as essential instruments in gauging whether novel medications surpass established therapies, thereby furnishing robust evidence to support their wider implementation.

This particular study stands out due to its core focus on the individual experiences of those confronting anorexia, actively engaged in a clinical trial incorporating medical interventions. The primary aim revolves around meticulously scrutinizing both trial

completion rates and instances of voluntary withdrawal within this specific patient cohort.

#### What are Observational Clinical Trials?

Participating in this medical trial involves engagement in an observational study, a pivotal aspect of clinical research meticulously crafted to glean insights through unobtrusive monitoring of patients as they adhere to their treatment protocols.

Researchers will simply observe your experience, meticulously assessing the outcomes of your condition without altering your treatment regimen. This trial design is instrumental in advancing our comprehension of the organic progression of a specific medical condition and its implications for individuals affected by it. Your voluntary involvement in this observational study contributes significantly to the advancement of medical knowledge and the refinement of care for individuals sharing the same ailment.

### Safeguarding Your Anonymity in the Research

Preserving the absolute confidentiality of your data remains a top priority throughout this study. To protect your anonymity, kindly avoid including any personal or identifiable details in your questionnaire responses. The dedicated research team is unwavering in their commitment to enhancing privacy and security measures. Nevertheless, it's important to acknowledge that certain legal circumstances may arise, compelling the disclosure of personal information.

## What Sets This Study Apart From Other Anorexia Clinical Trials

It is critical to recognize the unique character of this study endeavor. It is strictly observational, implying that your participation will not include particular therapies or interventions. Understanding the breadth of anorexia clinical research, including interventional studies incorporating various treatment regimens, is critical for making an educated decision regarding future involvement in a clinical trial.

Making an informed decision about future clinical trial participation necessitates an active strategy that includes research and trial comparison. Clinicaltrials.gov and other comparable websites include a plethora of information about <u>anorexia research</u>. In

addition, Power's specialized online platform provides a comprehensive list of ongoing anorexia clinical trials that are presently recruiting volunteers. With thorough research and a thorough understanding of the many clinical trial categories, you may safely select whether or not to enroll.

#### What You Need to Do

Your active participation is vital in this observational clinical study, where we encourage you to share your perspectives and experiences. This entails completing surveys every two weeks, taking approximately 20-30 minutes of your time. Additionally, our team is ready to conduct quarterly check-in calls to ensure ongoing support and your sustained engagement in the trial.

It's crucial to emphasize that your involvement in the survey phase of this trial is entirely voluntary. You have the autonomy to choose which questions to address or complete the entire questionnaire as per your discretion. Moreover, you retain the right to withdraw from the trial at any point. Recognizing the personal significance of participating in a clinical trial, our commitment lies in offering necessary support, respecting your privacy, and guiding your decision-making process throughout this trial.

# **Potential Advantages**

Participants in this observational clinical investigation may not experience immediate benefits; however, their involvement holds promise for long-term impact. The data collected from participants will contribute to the development of future approaches for engaging individuals coping with anorexia, potentially broadening horizons in medical research. Those engaged in this clinical trial have the potential to catalyze significant advancements in the field of medical research, potentially laying the groundwork for forthcoming anorexia patients.

#### Potential Health Outcomes and Hazards

Understanding potential health effects on participants, particularly in drug evaluation studies, remains crucial despite the advancements made through clinical trials.

However, in observational clinical research, we employ a distinct methodology to minimize these impacts by refraining from administering experimental medications to participants. Instead, our primary focus revolves around thorough monitoring and assessment of outcomes, guaranteeing the prevention of any avoidable health hazards.

## Facilitating Diversity in Clinical Studies

If you wish to delve into the complexities surrounding diversity within clinical trials, various online resources are available to deepen your understanding.

Whether your goal is to unravel the nuances of challenges and opportunities associated with diversity in clinical trials or expand your personal perspectives, these resources can serve as a valuable source of information:

Stewart, Jenell, Meighan L. Krows, Torin T. Schaafsma, Kate B. Heller, Elizabeth R. Brown, Jim Boonyaratanakornkit, Clare E. Brown et al. "Comparison of racial, ethnic, and geographic location diversity of participants enrolled in clinic-based vs 2 remote COVID-19 clinical trials." *JAMA Network Open* 5, no. 2 (2022): e2148325-e2148325.

Arieli, Daniella. "Emotional work and diversity in clinical placements of nursing students." *Journal of Nursing Scholarship* 45, no. 2 (2013): 192-201.

# Participant's Confirmation

I affirm that I've devoted ample time to grasp and internalize the contents of the informed consent form, either through individual review or with the guidance of professionals who elucidated its details. I'm pleased that all my queries have been satisfactorily addressed.

| Participant Name |
|-----------------------|
| Participant Signature |

| Date |
|---|
| Facilitator's Confirmation |
| I hereby confirm that I engaged in a comprehensive dialogue with the participant, meticulously explaining the intricacies contained within this written document. My objective was to ensure the participant's complete understanding of the primary research objectives, the methodology employed, potential risks and benefits, and other crucial elements of the anorexia clinical trial. |
| Printed Name of Assisting Researcher |
| Signature of Assisting Researcher |

Date